CLINICAL TRIAL: NCT05525104
Title: The Influence of Electroencephalographic Density Spectral Array Guidance of Sevoflurane Administration on Recovery From General Anaesthesia in Children Between 6 Months and 12 Years.
Brief Title: The Effect of DSA on Recovery of Anaesthesia in Children
Acronym: DSA-RCT-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Hannah Raab, BSc, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSA-RCT-1; NL80282.078.22 (Other: CCMO)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia; Depth of Hypnosis Monitoring
Keywords: Density spectral array; Depth of hypnosis; Paediatric anaesthesia

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and parents will be blinded to the treatment. The outcome assessor will be blinded as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): In patients randomised to the control group, sevoflurane will be titrated according to a Minimal Alveolar Concentration (MAC) of 0.9 respectively an end tidal sevoflurane concentration of 2.3% based on standard practice in our paediatric anaesthesia department.
- Treatment (Experimental): In patients randomised to the intervention group of the trial, the anaesthetic agent sevoflurane will be titrated according to the typical DSA pattern for general anaesthesia with sevoflurane, provided by the Narcotrend
  Interventions: Device: Narcotrend Monitor (MT MonitorTechnik, Hannover, Germany)

INTERVENTIONS:
Device: Narcotrend Monitor (MT MonitorTechnik, Hannover, Germany) — This trial is designed to investigate the additional value of Density Spectral Array monitoring, on the "speed of emergence" after general anaesthesia. We will compare traditional general anaesthesia with sevoflurane using a MAC value and subjective clinical parameters to the objective and continuous approach using DSA depth of hypnosis. The investigational product is the validated Narcotrend monitor, an electroencephalographic monitor, that is regularly used in anaesthesia practice in the Sophia children's hospital and will be used according to intended purpose. The extended version as used in the operating room in the Sophia Children's hospital offers a diversity of diagrams including Density Spectral Array.
  The electroencephalographic Narcotrend monitor records frontal EEG-activity. Standard paediatric ECG electrodes are used for EEG registration
  Arms: Treatment

SUMMARY:
In this randomised, blinded study, we will investigate the influence of DSA on recovery from general anaesthesia. DSA monitoring provides continuous information on depth of hypnosis. Based on DSA monitoring dose adjustments of sevoflurane can be made. We expect that this will lead to a faster speed of emergence and recovery.

DETAILED DESCRIPTION:
Electroencephalographic density spectral array (DSA) is a three dimensional method to display electroencephalogram (EEG) signals consisting of the EEG frequency (y-axis), the power of the EEG signal (colour-coded to be integrated into a two dimensional plot) and the development of the EEG power spectrum over time (x-axis). DSA is routinely used to measure depth of hypnosis (DoH) by a part of the staff members in our department. When DSA is used, dose adjustments of sevoflurane will be made based on monitoring depth of anaesthesia. However, most of our colleague do not use DSA. Dose adjustment is then based on (subjective) clinical surrogate parameters, or in general mostly based on a minimal alveolar concentration of the anaesthetic gas that is used.

Electroencephalographic DSA monitoring provides continuous objective information on DoH and should result in a faster speed of emergence and recovery from general anaesthesia (GA). This will be addressed in a randomised controlled trial.

In patients randomised to the intervention group, the anaesthetic agent sevoflurane will be administered on the basis of objective measures of anaesthetic depth, the typical DSA pattern for GA. We expect a significantly faster speed of emergence and recovery in the intervention group based on clinical experience. The Narcotrend monitor is validated for use in paediatric patients. There are thus no additional risk factors apart from those, which are inherent with general anaesthesia. Patient randomised to the control group will receive standard treatment, that is delivery of sevoflurane based on a MAC of 0.9 respectively an end tidal sevoflurane concentration of 2.3%. A non-invasive therapeutical intervention (DSA based conduct of GA) should result in the advantage of faster recovery, without any additional risk factor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of parents/guardians
* Age ≥6 months and ≤12 years
* Surgical procedure requiring GA supplemented with caudal analgesia
* Ability of the parents/guardians to communicate in Dutch

Exclusion Criteria:

* Primary exclusion criteria
* Withdrawal of informed consent
* (Chronic) use of drugs influencing the electroencephalogram
* Use of premedication
* Known intolerance for sevoflurane
* Parents/guardians unable to communicate in Dutch
* Secondary exclusion criteria
* Protocol violation
* Data registration failure

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Weber, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data of a patient will only be shared with other fellow researchers (e.g. in case of follow-up studies) upon reasonable request, on the condition that the child's parent explicitly consented.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available after data collection has been completed.
Access Criteria: Reasonable request of fellow researches and only data of patients after explicit consent from parents on the ICF.

REFERENCES:
- [Derived] de Heer IJ, Raab HAC, de Vries J, Karaoz-Bulut G, Weber F. The Influence of Electroencephalographic Density Spectral Array Guidance of Sevoflurane Administration on Recovery From General Anesthesia in Children. A Randomized Controlled Trial. Paediatr Anaesth. 2025 Apr;35(4):287-293. doi: 10.1111/pan.15065. Epub 2025 Jan 13. PMID 39803999

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: In patients randomised to the intervention group of the trial, the anaesthetic agent sevoflurane will be titrated according to the typical DSA pattern for general anaesthesia with sevoflurane, provided by the Narcotrend
  Narcotrend Monitor (MT MonitorTechnik, Hannover, Germany): This trial is designed to investigate the additional value of Density Spectral Array monitoring, on the "speed of emergence" after general anaesthesia. We will compare traditional general anaesthesia with sevoflurane using a MAC value and subjective clinical parameters to the objective and continuous approach using DSA depth of hypnosis. The investigational product is the validated Narcotrend monitor, an electroencephalographic monitor, that is regularly used in anaesthesia practice in the Sophia children's hospital and will be used according to intended purpose. The extended version as used in the operating room in the Sophia Children's hospital offers a diversity of diagrams including Density Spectral Array.
  The electroencephalographic Narcotrend monitor records frontal EEG-activity. Standard paediatric ECG electrodes are used for EEG registration
Period: Overall Study
Arm/Group | Control | Treatment
Started | 56 | 56
Completed | 44 | 52
Not Completed | 12 | 4
Not completed — Failed caudal analgesia | 1 | 3
Not completed — Premedication needed | 0 | 1
Not completed — Protocol Violation | 10 | 0
Not completed — Cancelled operation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 44 | 52 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.2 (2.6) | 2.4 (2.7) | 2.3 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 40 | 48 | 88
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kilogram] | 13.6 (6.3) | 13.8 (6.6) | 13.7 (6.4)
ASA-score [Count of Participants; unit: Participants] — The ASA classification is a system to assess and communicate a patient's pre-anesthesia medical co-morbidities. It ranges from 1 to 6. An ASA-classification of 1 equals a healthy patient, 2 equals mild systemic disease (e.g. asthma without exacerbation) and 3 severe systemic disease (e.g. asthma with exacerbation). Along with other risk factors, it can be used to predict perioperative risks.
  Participants
    1 | 37 | 46 | 83
    2 | 6 | 6 | 12
    3 | 1 | 0 | 1
Type of surgery [Count of Participants; unit: Participants]
  Orchidopexy | 18 | 15 | 33
  Inguinal hernia repair | 9 | 8 | 17
  Urethral valves repair | 0 | 1 | 1
  Hypospadias correction | 9 | 13 | 22
  Cystoscopy/Sachse or meatotomy | 3 | 11 | 14
  Other urological | 4 | 4 | 8
  Orthopedic surgery | 1 | 0 | 1
Duration of general anesthesia [Mean (Standard Deviation); unit: minutes] | 83.7 (39.1) | 69.4 (37.2) | 75.5 (36.8)

OUTCOME MEASURES:

1. Primary Outcome: The Influence of DSA Monitoring on the Speed of Emergence.
Description: The speed of emergence is defined as the time interval between the end of hypnotic drug application and the moment when discharge criteria from the operating room are met (defined as a Steward score ≥ 3)
  The Steward recovery score consists of three domains: consciousness, airway and motor. Consciousness can be scored from 0-2, in which 0 equals non responsive, 1 equals response to stimuli, 2 equals awake. Airway is scored from 0-2: airway that requires maintenance scores 0, maintaining good airway scores 1 and coughing on command or crying scores 2. Motor is also scored form 0-2: no movement scores 0, non-purposeful movement scores 1 and purposeful movement scores 2. Combining all three domains, the minimum score is 0 (unconscious) and the maximum score is 6 (completely awake) The speed of emergence is defined as a minimum score of 3, with a minimum score of 1 in each domain.
Time Frame: Day 0
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Control | Treatment
Number analyzed (Participants) | 44 | 52
minutes | 12 [6 to 24.3] | 6 [4 to 16.8]
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.041, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Total Time From Discontinuation of Anaesthetic Drug Delivery Until Discharge From the Post Anaesthesia Care Unit.
Description: The total time is defined as the time interval between the end of hypnotic drug application and the moment when discharge criteria from the recovery room are met (defined as a Steward score =6)
  The Steward recovery score consists of three domains: consciousness, airway and motor. Consciousness can be scored from 0-2, in which 0 equals non responsive, 1 equals response to stimuli, 2 equals awake. Airway is scored from 0-2: airway that requires maintenance scores 0, maintaining good airway scores 1 and coughing on command or crying scores 2. Motor is also scored form 0-2: no movement scores 0, non-purposeful movement scores 1 and purposeful movement scores 2. Combining all three domains, the minimum score is 0 (unconscious) and the maximum score is 6 (completely awake).
Time Frame: Day 0
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Control | Treatment
Number analyzed (Participants) | 44 | 52
minutes | 26.5 [12.3 to 40.5] | 18.5 [7 to 32.5]
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.066, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: The Incidence of Postoperative Delirium
Description: The incidence of postoperative delirium is assessed with the Cornell assessment of postoperative delirium (is defined as a score equal to or greater than 9).
  The Cornell assessment of postoperative delirium consists of eight questions. The first four questions are scored as follows: 0 equals always, 1 often, 2 sometimes, 3 rarely, 4 never.
  1. Does the child make eye contact with the caregiver?
  2. Are the child's actions purposeful?
  3. Is the child aware of his/her surroundings?
  4. Does the child communicatie needs and wants? In these first four questions, a higher score represents a worse outcome.
     The last four questions are scored as follows: 0 equals never, 1 rarely, 2 sometimes, 3 often and 4 always.
  5. Is the child restless?
  6. Is the child inconsolable?
  7. Is the child underactive - very little movement while awake?
  8. Does it take the child a long time to respond to interactions? In these last four questions, a higher score represents a worse outcome.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 44 | 52
Participants | 0 | 0

4. Secondary Outcome: Differences of Depth of Hypnosis During the Procedure, as Measured by the Narcotrend Monitor.
Description: Density spectral array patterns will be saved, and divided into categories, which will be compared between the two study groups.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 44 | 52
Participants
  DSA pattern representing general anesthesia | 24 | 46
  DSA pattern representing too deep anesthesia | 20 | 4
  DSA pattern representing lighter anesthesia | 0 | 2

5. Secondary Outcome: Incidence of Recall of Events During the Procedure (Awareness)
Description: Awareness is assessed with a modified Brice interview in children of 6 years or older.
Time Frame: Day 0, Day 1, Day 14
Population: Interviews only conducted in children ≥6 years
Measure: Number; unit: participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 6 | 7
participants
  Day 0 | 0 | 0
  Day 1 | 0 | 0
  Day 14 | 0 | 0

6. Secondary Outcome: The End-tidal Sevoflurane Concentration
Description: The mean end-tidal sevoflurane concentration measured during surgical procedure
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: percentage sevoflurane of exhaled air
Arm/Group | Control | Treatment
Number analyzed (Participants) | 44 | 52
percentage sevoflurane of exhaled air | 2.3 (0.1) | 1.8 (0.34)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the entire study period: until the patiënt was discharged (on average 3-6 hours after anesthesia) or until the last Brice interview was conducted if the patient was 6 years or older (2 weeks after anesthesia).
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/52
Other Adverse Events (participants affected / at risk) | 3/44 | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=44) | Treatment (N=52)
Prolonged hospitalisation (Infections and infestations) | 0 (0) | 1 (1) — The surgery was performed in day care, but the patient required longer hospitalization due to underlying disease (not related to anesthesia or study participation)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=44) | Treatment (N=52)
Decrease in blood pressure (-2 SD) (Cardiac disorders) | 3 (3) | 0 (0) — A decrease in blood pressure (of -2 SD) that could be remedied with an intravenous fluid bolus which had no further consequences for the patient.

LIMITATIONS AND CAVEATS:
The relatively large number of secondary exclusions due to protocol violations in the standard care group is a shortcoming of this study. The target number of 51 participants per study group was not achieved. Because this exclusion due to protocol violation is completely patient independent, confounding due to exclusion for an outcome-related reason is not an issue. So, to identify a treatment effect that would occur under optimal conditions, we choose to perform a per-protocol analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT05525104/Prot_SAP_000.pdf